CLINICAL TRIAL: NCT06124183
Title: Results of an Emotional Intelligence Program for Adolescent Offenders Based on Salovey and Mayer's Ability Model.
Brief Title: Emotional Intelligence Program for Adolescents With Antisocial Behavior (DYNAMIS)
Acronym: DYNAMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Valle, Colombia (Other)
Collaborators: Universidad de la Sabana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1102812; PSI2017-84005-R (Other Grant/Funding Number: Spanish Ministry of Science, Innovation and Universities)
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-01

CONDITIONS: Mental Health Wellness 1
Keywords: Depression; Anxiety; Stress; Emotions; Subjective well-being
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The design was a quasi-experimental study with intervention and control groups and pre-post-intervention measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): A 12-session psychological program The intervention program consisted of 12 sessions of 80 minutes with a weekly frequency. The first session was diagnostic, and the following nine correspond to the following topics: perception (2), facilitation (2), labeling and understanding (2), emotional regulation, and management (3). The last session was evaluative. The intervention included practical tasks in context and supervision by clinical psychologist.
  Interventions: Behavioral: The program comprises 12 sessions and additional activities to be carried out after each session, alongside counseling from the program's leading professionals
- Control Group (Placebo Comparator): Does not receive intervention
  Interventions: Behavioral: The program comprises 12 sessions and additional activities to be carried out after each session, alongside counseling from the program's leading professionals

INTERVENTIONS:
Behavioral: The program comprises 12 sessions and additional activities to be carried out after each session, alongside counseling from the program's leading professionals — The program is based on the emotional intelligence skills model (Mayer & Salovey, 1997; Salovey & Mayer, 1990), which suggests that emotional intelligence consists of four hierarchical branches or components: (a) perception of emotions, (b) facilitating thinking using emotions, (c) understanding emotions, and (d) managing and handling emotions. The program comprises 12 sessions and additional activities to be carried out after each session, alongside counseling from the program's leading professionals. The sessions follow a similar structure, involving session framing, motivation on the central theme, group activity for sharing ideas and experiences, individual activities, review, and task assignment. The first and second sections focus on analyzing the personal reality and current emotional conditions of the participants, while the final session is designed for both celebration and program evaluation. The remaining nine sessions address the four branches of the skill model.

SUMMARY:
This study assessed the effectiveness of an emotional intelligence program based on the Salovey and Mayer model among adolescents exhibiting antisocial behavior. A quasi-experimental design was employed, involving 231 Colombian adolescent offenders (122 in the experimental group). A 12-session psychological protocol was implemented. The primary question it aims to address is whether it is feasible for adolescents with antisocial behavior to reduce negative emotional symptoms related to mental health, such as anxiety, stress, and depression, while simultaneously improving their emotional skills. It was observed that those who completed the program showed significant improvements in emotional intelligence, emotional balance, and resilience while experiencing a decrease in emotional symptoms, particularly in stress.

DETAILED DESCRIPTION:
Emotional intelligence programs have been shown to enhance mental health, social adjustment, and overall well-being in adolescents, primarily implemented in educational settings but adaptable to specific clinical populations. The goal of this study was to assess the effectiveness of an emotional intelligence program tailored for adolescents with antisocial behavior based on the Salovey and Mayer ability model. Given previous findings suggesting that emotional intelligence programs can aid in improving mental health and social adjustment in adolescents, there arises a need to evaluate the efficacy of such programs in correctional settings. This study aimed to ascertain the effectiveness of an emotional intelligence program designed for adolescents with antisocial behavior. It also supported the notion that implementing emotional intelligence programs in socio-educational centers working with such adolescents could be an effective strategy to enhance their psychological and social well-being. Additionally, it highlights the necessity of incorporating emotional intelligence training in intervention processes within correctional contexts.

The study employed a quasi-experimental design with both intervention and control groups, conducting pre-post intervention measures. The study involved 231 Colombian adolescent participants aged between 14 and 18 (Mean = 15.55, SD = 1.30), with 122 in the intervention group (Mean = 15.64, SD = 1.29, 19.7% female) and 109 in the control group (Mean = 15.44, SD = 1.30, 27.5% female). Questionnaires were utilized to evaluate emotional intelligence, emotional experiences, resilience, emotional symptoms (depression, anxiety, and stress), and life satisfaction.

The comparative analyses revealed significant differences between the intervention and control groups. Adolescents who completed the program demonstrated improvements in emotional intelligence, emotional balance, and resilience while experiencing a notable reduction in emotional symptoms, particularly stress.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were being enrolled in the first year or higher grades of secondary education, having parental and authority permission, and being between 14 and 18 years old

Exclusion Criteria:

* The exclusion criteria were being younger than 14 or older than 18, openly refusing to participate, lacking authorization, and having the scheduled completion of the judicial measure during the program execution period.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants were asked which gender they identified with.
Enrollment: 231 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Emotional Intelligence | 4 months
  Attention, Clarity and Emotional Repair. Trait Meta Mood Scale (TMMS-24)
Emotional Intelligence | 4 months. It offers five alternative answers. High scores on the factors indicate a higher degree of emotional intelligence.
  Attention, Clarity and Emotional Repair. Trait Meta Mood Scale (TMMS-24)
Emotional symptoms of mental health | 4 months. The scale rates emotional symptoms from normal to extremely severe. Depression (0-9, normal- 28+ extremely severe). Anxiety (0-7, normal- 20+ extremely severe). Stress (0-4, normal- 34+ extremely severe.
  Depression, anxiety and stress scale (DASS-21)
Positive and negative emotional experiences | 4 months. The items are presented on a Likert scale ranging from "Very rarely or never" to "Very often or always" (5).(Range 5-30)
  Positive and negative emotional experiences (SPANE)

SECONDARY OUTCOMES:
Affective balance | 4 months. The affective balance scale is derived from the difference between the two SPANE sub-scales (SPANE-P and SPANE-N).
  Positive and negative emotional experiences scale (SPANE)
Satisfaction with life | 4 months. Scores between 31-35 indicate the individual is very satisfied; 26-30, satisfied; 21-25, somewhat satisfied; 20, neutral; 15-19, somewhat dissatisfied; 10-14, dissatisfied; and 5-9, very dissatisfied.
  Satisfaction with life Scale (SWLS)
Resilience | 4 months. It consists of 10 items designed as a Likert-type scale with five response options. The final score for the questionnaire is obtained by summing the responses (range 0-40).
  Connor-Davidson Resilience Scale (CD-RISC-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Arcadio de Jesús Cardona Isaza, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available whit request to the authors.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: Undefined
Access Criteria: The data that support the findings of this study are available whit request to the authors.